CLINICAL TRIAL: NCT00636961
Title: An Exploratory, Double Blind, Randomized, Placebo-controlled, 2-way Cross-over Study to Assess the Effect of Repeat-dose Inhaled Indacaterol Maleate (300 μg) on Dynamic and Static Lung Hyperinflation, Subjective Breathlessness and Health Status in Patients With COPD
Brief Title: An Exploratory Study, to Assess the Effect of Repeat-dose Inhaled Indacaterol Maleate (300 μg) on Dynamic and Static Lung Hyperinflation, Subjective Breathlessness and Health Status in Patients With Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CQAB149B2318
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Indacaterol Maleate, Exercise testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: Indacaterol 300μg followed by Placebo (Experimental): In period I, indacaterol 300μg was taken by inhalation once daily via the Concept 1 inhaler device for 2 weeks. In period II, matching placebo was taken by inhalation once daily via the Concept 1 inhaler device for 2 weeks. For each treatment period and for each patient, the doses were to be administered between 7am and 12am. A period of at least 4 days but no more than 21 days separated each treatment period. Rescue medication (short-acting beta-agonist (SABA)) was prescribed by the investigator for the duration of the study.
  Interventions: Drug: Indacaterol 300μg; Drug: Placebo
- Sequence 2 : Placebo followed by Indacaterol 300μg (Experimental): In period I, matching placebo was taken by inhalation once daily via the Concept 1 inhaler device for 2 weeks. In period II, indacaterol 300μg was taken by inhalation once daily via the Concept 1 inhaler device for 2 weeks. For each treatment period and for each patient, the doses were to be administered between 7am and 12am. A period of at least 4 days but no more than 21 days separated each treatment period. Rescue medication (short-acting beta-agonist (SABA)) was prescribed by the investigator for the duration of the study.
  Interventions: Drug: Indacaterol 300μg; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol 300μg — 300μg indacaterol maleate inhalation powder in hard gelatin capsules administered via Concept1 inhalation device
  Other Names: Arcapta
Drug: Placebo — Matching placebo devices and hard gelatin capsules

SUMMARY:
This study evaluated the effect of QAB149 on dynamic and static hyperinflation, breathlessness, and health status in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects,
* 40 to 80 years of age,
* with a documented diagnosis of mild, moderate or severe chronic obstructive pulmonary disease (COPD) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria and >20-pack year history of smoking, a post-bronchodilator 40% ≤ FEV1 ≤ 80% of predicted normal and post-bronchodilator FEV1/FVC < 70% who have signed an informed consent form (ICF) prior to the initiation of any study-related procedure (Post bronchodilator refers to 30 minutes after the inhalation of 400 µg of salbutamol)
* Subjects who demonstrate a plethysmographic functional residual capacity >120% predicted normal

Exclusion Criteria:

* No COPD exacerbations within 6 weeks prior to dosing,
* no concomitant lung disease such as asthma,
* no requirement for long term oxygen treatment or history of lung reduction surgery.
* No medical conditions that would interfere with the performance of spirometry or clinical exercise testing.
* Any other medical condition that in the opinion of the investigator may cause the patient to be unsuitable for completion of the study or place the patient at potential risk from participating in the study e.g. uncontrolled hypertension or unstable ischemic heart disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (3):
- Germany (3):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Mönchengladbach
  - Novartis Investigator Site, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Sequence 1: Indacaterol 300μg Followed by Placebo | Sequence 2 : Placebo Followed by Indacaterol 300μg
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1
Not completed — Administrative problems | 1 | 1
Period: Period 2
Arm/Group | Sequence 1: Indacaterol 300μg Followed by Placebo | Sequence 2 : Placebo Followed by Indacaterol 300μg
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Indacaterol 300μg Followed by Placebo | Sequence 2 : Placebo Followed by Indacaterol 300μg | Total
Number analyzed (Participants) | 14 | 13 | 27
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measurements are based on total randomized patients.
  years | 62.6 (8.30) | 59.8 (5.81) | 61.3 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Capacity (IC) at Peak Time and at Isotime on Day 14
Description: Inspiratory capacity (IC) at peak time and at isotime were the primary pharmacodynamic (PD) variables of interest. IC was measured at two minute intervals during exercise. Isotime was defined as the time the subject was still exercising in the shortest of all sub-maximal exercise tests (3-minutes resting pedaling, 3-minutes unloaded pedaling and exercise with loaded pedaling). Peak time was defined as the last measurement taken in the exercise period. The primary analysis consisted of a linear mixed effects model with baseline IC measurement as covariate.
Time Frame: Day 14
Population: The safety analysis set consisted of all patients who received study medication and had at least one assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Groups:
- Indacaterol 300ug: Patients received indacaterol 300μg via the Concept 1 inhaler device once daily (between 7 am and 12 am) for 2 weeks. Rescue medication (SABA) was prescribed by the investigator for the duration of the study.
- Placebo: Patients received matching placebo via the Concept 1 inhaler device once daily in the morning (between 7 am to 12am) for 2 weeks. Rescue medication (SABA) was prescribed by the investigator for the duration of the study.
Arm/Group | Indacaterol 300ug | Placebo
Number analyzed (Participants) | 25 | 25
Liters
  IC at Peak | 2.36 [2.25 to 2.48] | 2.05 [1.93 to 2.16]
  IC at Isotime | 2.37 [2.25 to 2.48] | 2.10 [1.99 to 2.21]

2. Secondary Outcome: Static Inspiratory Capacity (IC) at Day 14
Description: Inspiratory Capacity (IC) at resting (static IC) was measured by using whole body plethysmography. The day 14 measurement was analyzed using an analysis of variance including baseline (day -2) as a covariate,
Time Frame: Day 14
Population: The safety analysis set consisted of all patients who received study medication and had at least one assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 300ug | Placebo
Number analyzed (Participants) | 26 | 26
Liters | 2.55 [2.46 to 2.65] | 2.37 [2.28 to 2.47]

3. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Measured by Spirometry on Day 14
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose. The linear mixed model included the baseline FEV1 measurement as covariate.
Time Frame: Day 14
Population: The safety analysis set consisted of all patients who received study medication and had at least one assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 300ug | Placebo
Number analyzed (Participants) | 25 | 25
Liters | 1.68 [1.59 to 1.76] | 1.53 [1.45 to 1.62]

4. Secondary Outcome: Chronic Activity Related Breathlessness Measured by Transition Dyspnoea Index (TDI) at Day 14
Description: Dyspnoea was measured during the treatment period using the transition dyspnoea index (TDI), which captures changes from baseline. The TDI has three domains; functional impairment, magnitude of task and magnitude of effort. TDI domains are rated from -3 (major deterioration) to 3 (major improvement) and rates are summed for transition focal score ranging from -9 to 9; minus scores indicate deterioration. A TDI focal score of 1 was considered to be a clinically significant and meaningful improvement from baseline. Analysis of variance included period baseline dyspnoea index (BDI) as covariate.
Time Frame: Day 14
Population: The safety analysis set consisted of all patients who received study medication and had at least one assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score on a scale
Arm/Group | Indacaterol 300ug | Placebo
Number analyzed (Participants) | 20 | 22
Score on a scale | 1.0 [-0.3 to 2.4] | -2.3 [-3.6 to -1.0]

5. Secondary Outcome: Dyspnoea Measured by Borg CR10 Scale at Day 1, Day 14
Description: The modified Borg CR10 Scale consists of 12-point score that the patients point to so as to indicate their level of dyspnoea (where 0 indicates no breathlessness at all to 12 indicates maximum breathlessness), before and during exercise testing. A reduction in this score indicates an improvement. Isotime was defined as the time the subject was still exercising in the shortest of all sub-maximal exercise tests. Peak time was defined as the last measurement taken in the exercise period. Analysis of variance included period, treatment and sequence as fixed effects and subject as random effect.
Time Frame: Day 1, Day 14
Population: The safety analysis set consisted of all patients who received study medication and had at least one assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score on a scale
Arm/Group | Indacaterol 300ug | Placebo
Number analyzed (Participants) | 26 | 26
Score on a scale
  Day 1 : score at Peak (n= 26, 26) | 8.2 [7.4 to 8.9] | 7.9 [7.2 to 8.7]
  Day 14: score at Peak (n= 25, 25) | 8.1 [7.5 to 8.8] | 8.7 [8.1 to 9.4]
  Day 1 : score at Isotime (n= 26, 26) | 5.9 [5.0 to 6.7] | 5.8 [4.9 to 6.6]
  Day 14 : score at Isotime(n= 25, 25) | 5.2 [4.4 to 6.0] | 6.7 [5.9 to 7.5]

ADVERSE EVENTS:
Description: The safety analysis set that consisted of all patients who received study medication and had at least one assessment.
Arm/Group | Indacaterol 300ug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 9/26 | 9/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300ug (N=26) | Placebo (N=26)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.